CLINICAL TRIAL: NCT01967433
Title: Use of Diphenhydramine as an Adjunctive Sedative for Colonoscopy in Patients Chronically on Opioids
Brief Title: Diphenhydramine as an Adjunctive Sedative in Patients on Chronic Opioids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DAASIPCO
Record Dates: First submitted 2013-10-11; First posted 2013-10-22 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Colonoscopy; Adjunct Anesthesia Medication
Keywords: Fentanyl; Midazolam; Sedation; Patient tolerance; Duration of colonoscopy
MeSH Terms: interventions — Diphenhydramine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diphenhydramine (Experimental): Diphenhydramine 50 mg IV 3 minutes prior to administration of other sedatives
  Interventions: Drug: Diphenhydramine
- Placebo (Placebo Comparator): 0.9% sodium chloride 10 ml IV 3 minuted prior to administration of other sedatives
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diphenhydramine
  Other Names: Benadryl
  Arms: Diphenhydramine
Drug: Placebo
  Other Names: Normal Saline; 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
To access the efficacy of adding diphenhydramine as adjunct to improve sedation and to reduce the amount of standard sedatives used during colonoscopy in patients on chronic opioids.

DETAILED DESCRIPTION:
Specific Aims:

The primary aim of our study is to determine if addition of Diphenhydramine to Fentanyl and Midazolam will decrease the dose of Fentanyl and Midazolam used during colonoscopy in individuals on chronic opioids. Secondarily we will be looking at quality of sedation, duration of colonoscopy, time to reach cecum and adverse effects (hypoxia defined as O2 saturation less than 89% lasting for more than 30 seconds, hypotension defined as systolic BP less than 90 mmhg and use of reversal agents i.e Naloxone or Flumazenil).

Day of Procedure:

After consent is obtained the medical records of the patients will be reviewed and demographic information, co-morbidities, current medication will be extracted and recorded.

On the day of colonoscopy Alcohol use disorder inventory (AUDIT) will be used to screen for alcohol abuse. AUDIT was developed by World Health Organization and has been validated over a period of 2 decades. It consist of 10 questions, each question is scored 0-4 on the basis of subjects alcohol use. It takes about 2-4 minutes to complete. A score 10 or greater is highly specific or alcohol use.

Subjects will be checked in and prepared according to routine protocols of the VA medical center. Participants will be randomly assigned to receive either 50 mg of diphenhydramine or 10 ml of 0.9% sodium chloride. On the day of colonoscopy randomization will be performed by an independent investigator who is a pharmacist at VA medical center using the website http://www.randomization.com. She will also prepare and dispense medication. Each endoscopy team will consist of an attending gastroenterologist, gastroenterology fellow and two nurses. Medications will be administered by one of the nurses under the direct supervision of the physician.

At the start of procedure baseline vitals will be recorded as per our unit's policy. Research medication will be administered 3 minutes prior to administration of other medications. Neither the patient nor the medical staff including the endoscopist will be aware of the contents of the vial. Conscious sedation will be achieved using a combination of intravenous midazolam and fentanyl as standard sedative. Rarely, additional diphenhydramine will be given, on the basis of the judgment of the endoscopist. During the procedure vital signs including oxygen saturation will be monitored at 3-5 minute interval. Procedure related complications, including hypotension, desaturation and cardiac arrhythmia will be managed according to our endoscopy unit policy and protocols.

Following the procedure, the nurse and the fellow or the attending will individually rate the quality if sedation on a ten-point Likert scale. Qualitative assessment will also be made (Under-sedated, adequately sedated, or over-sedated).

Recovery time will be recorded.

Day Following the Colonoscopy Twenty-four hour discharge a follow up call will be made and the patients will be asked to evaluate the level of sedation on a 10-point scale (1, inadequate; 10 completely without discomfort); pain (1, no pain; 10 severe pain), and amnesia (10, no memory of the procedure; 1 complete memory).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-64 years undergoing screening, surveillance, diagnostic and therapeutic colonoscopy
* Patient on chronic opioids defined as at least 5 mg of morphine or its equivalent at least 3 days per week for more than 3 months

Exclusion Criteria:

* Inability to execute informed consent
* Allergy to Diphenhydramine, fentanyl or midazolam
* Known or suspected pregnancy
* Endoscopic procedure without sedation
* Patient scheduled to have other endoscopic procedures on the same day
* Prior alimentary tract surgery
* Severe cardiopulmonary disease (ASA IV)
* Monoamine Oxidase Inhibitors (MOI) use within 2 weeks of procedure

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-12; Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salman Nusrat, MD, Study Director — University of Oklahoma; Mohammad Madhoun, MD MS, Principal Investigator — Univeristy of Oklahoma Health Sciences Center
Locations (1):
- Veterans Affairs Medical Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Abraham NS, Fallone CA, Mayrand S, Huang J, Wieczorek P, Barkun AN. Sedation versus no sedation in the performance of diagnostic upper gastrointestinal endoscopy: a Canadian randomized controlled cost-outcome study. Am J Gastroenterol. 2004 Sep;99(9):1692-9. doi: 10.1111/j.1572-0241.2004.40157.x. PMID 15330904
- [Background] Zubarik R, Ganguly E, Benway D, Ferrentino N, Moses P, Vecchio J. Procedure-related abdominal discomfort in patients undergoing colorectal cancer screening: a comparison of colonoscopy and flexible sigmoidoscopy. Am J Gastroenterol. 2002 Dec;97(12):3056-61. doi: 10.1111/j.1572-0241.2002.07101.x. PMID 12492190
- [Background] Bergeron P, Enns J, Delima L, Dupuis JY, Wynands JE. Effects of routine premedication for cardiac catheterization on sedation, level of anxiety and arterial oxygen saturation. Can J Cardiol. 1995 Mar;11(3):201-5. PMID 7889437
- [Background] Cook PJ, Flanagan R, James IM. Diazepam tolerance: effect of age, regular sedation, and alcohol. Br Med J (Clin Res Ed). 1984 Aug 11;289(6441):351-3. doi: 10.1136/bmj.289.6441.351. PMID 6432093
- [Background] Pena LR, Mardini HE, Nickl NJ. Development of an instrument to assess and predict satisfaction and poor tolerance among patients undergoing endoscopic procedures. Dig Dis Sci. 2005 Oct;50(10):1860-71. doi: 10.1007/s10620-005-2952-7. PMID 16187188
- [Background] Keeffe EB, O'Connor KW. 1989 A/S/G/E survey of endoscopic sedation and monitoring practices. Gastrointest Endosc. 1990 May-Jun;36(3 Suppl):S13-8. PMID 2351253
- [Background] Hirsh I, Vaissler A, Chernin J, Segol O, Pizov R. Fentanyl or tramadol, with midazolam, for outpatient colonoscopy: analgesia, sedation, and safety. Dig Dis Sci. 2006 Nov;51(11):1946-51. doi: 10.1007/s10620-006-9413-9. Epub 2006 Sep 29. PMID 17009113
- [Background] Tu RH, Grewall P, Leung JW, Suryaprasad AG, Sheykhzadeh PI, Doan C, Garcia JC, Zhang N, Prindiville T, Mann S, Trudeau W. Diphenhydramine as an adjunct to sedation for colonoscopy: a double-blind randomized, placebo-controlled study. Gastrointest Endosc. 2006 Jan;63(1):87-94. doi: 10.1016/j.gie.2005.08.015. PMID 16377322
- [Background] Roach CL, Husain N, Zabinsky J, Welch E, Garg R. Moderate sedation for echocardiography of preschoolers. Pediatr Cardiol. 2010 May;31(4):469-73. doi: 10.1007/s00246-009-9622-z. Epub 2010 Jan 3. PMID 20047024
- [Background] Hofmeister EH, Egger CM. Evaluation of diphenhydramine as a sedative for dogs. J Am Vet Med Assoc. 2005 Apr 1;226(7):1092-4. doi: 10.2460/javma.2005.226.1092. PMID 15825733
- [Background] Husain Z, Hussain K, Nair R, Steinman R. Diphenhydramine induced QT prolongation and torsade de pointes: An uncommon effect of a common drug. Cardiol J. 2010;17(5):509-11. PMID 20865683

RESULTS

PARTICIPANT FLOW:
Groups:
- Diphenhydramine: Diphenhydramine 50 mg IV 3 minutes prior to administration of other sedatives
  Diphenhydramine Allocated: 61 Lost to follow up: 0 Analyzed: 61
- Placebo: 0.9% sodium chloride 10 ml IV 3 minuted prior to administration of other sedatives
  Placebo Allocated: 59 Lost to follow up: 0 Analyzed: 58
Period: Overall Study
Arm/Group | Diphenhydramine | Placebo
Started | 61 | 59
Completed | 61 | 58
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diphenhydramine | Placebo | Total
Number analyzed (Participants) | 61 | 58 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.3) | 60.1 (9.7) | 60.37 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 57 | 56 | 113
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 45 | 46 | 91
  Race: Others | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 61 | 58 | 119

OUTCOME MEASURES:

1. Primary Outcome: Dosage of Fentanyl
Description: Moderate sedation (using the American Society of Anesthesiologists definition of maintaining purposeful response to verbal or tactile stimulation, adequate ventilation requiring no airway protection, and maintenance of cardiovascular function) was then achieved using incremental doses of the combination of intravenous midazolam (1 mg) and fentanyl (25 μg) given every 2 to 3 minutes. To minimize any crossover, additional diphenhydramine was not permitted.
Time Frame: From induction (first dose of sedative) to end of procedure
Measure: Mean (Standard Deviation); unit: (μg)
Groups:
- Diphenhydramine: Diphenhydramine 50 mg IV 3 minutes prior to administration of other sedatives
  Diphenhydramine
- Placebo: 0.9% sodium chloride 10 ml IV 3 minuted prior to administration of other sedatives
  Placebo
Arm/Group | Diphenhydramine | Placebo
Number analyzed (Participants) | 61 | 58
(μg) | 125.4 (56.2) | 126.9 (53.5)

2. Secondary Outcome: Quality of Sedation
Description: Quality of sedation will be accessed by the nurse and the physician at the end of procedure.
  Name: 10 point visual analogue scale Minimum score: 1 (worse) Maximum score: 10 (better)
Time Frame: During the colonoscopy and 24 hours after discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diphenhydramine | Placebo
Number analyzed (Participants) | 61 | 58
score on a scale
  Physician rating | 6.2 (1.1) | 5.3 (1.2)
  Nurse rating | 5.6 (1.5) | 5.1 (1.4)

3. Secondary Outcome: Duration of Procedure
Description: Induction period (time from first dose of fentanyl to scope insertion), procedural time (time from scope insertion to scope out), and recovery time (time from scope out to discharge) were recorded by the nursing staff in their standard documentation.
Time Frame: Time from induction (first dose of sedative) to discharge
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Diphenhydramine | Placebo
Number analyzed (Participants) | 61 | 58
minutes
  Procedure time | 34.8 (19.5) | 34.7 (17.8)
  Recovery | 34.4 (9.2) | 32.4 (5.9)
  Induction | 6.4 (3.2) | 6.3 (2.8)

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Following adverse events will be recorded: (1)Hypoxia defined as O2 saturation less than 89% lasting for more than 30 seconds, (2)hypotension defined as systolic BP less than 90 mmhg and (3)use of reversal agents i.e Naloxone or Flumazenil
Time Frame: From induction (first dose of sedative) to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Diphenhydramine | Placebo
Number analyzed (Participants) | 61 | 58
Participants
  Hypotension | 12 | 22
  Hypertension | 5 | 3
  Desaturation | 0 | 0
  Apnea | 0 | 0
  Arrhythmia | 0 | 0
  Reversal agent use | 0 | 0
  Tachypnea | 0 | 0

5. Secondary Outcome: 24 Hour Follow up Pain Score
Description: At 24 hr follow up patients were asked to rate the level of pain during the procedure using 10 point scale.
  10 point visual analogue scale minimum= 0 (better) maximum =10 (worse)
Time Frame: About 24 hours after the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diphenhydramine | Placebo
Number analyzed (Participants) | 61 | 58
score on a scale | 2.0 (2.17) | 3.09 (3.95)

6. Secondary Outcome: Dosage of Midazolam
Description: as for outcome 1
Time Frame: From induction (first dose of sedative) to end of procedure
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Diphenhydramine | Placebo
Number analyzed (Participants) | 61 | 58
mg | 4.9 (2.1) | 5.0 (1.9)

7. Secondary Outcome: 24 Hour Follow up Amnesia Score
Description: Patient were also asked to rate amnesia on a 10 point scale 24 after discharge. minimum= 0 (worse) maximum =10 (better)
Time Frame: At about 24 after the procedure
Measure: Mean (Standard Deviation); unit: score on a 10 point point scale
Arm/Group | Placebo | Diphenhydramine
Number analyzed (Participants) | 61 | 58
score on a 10 point point scale | 7.8 (3.4) | 6.5 (3.8)

ADVERSE EVENTS:
Time Frame: Preprocedure, procedural, post procedure and 24 hr follow up
Description: Hypoxia (defined as O 2 saturation less than 89% lasting for more than 30 seconds), hypertension (20 mm Hg increase in blood pressure from baseline, provided this is >140 mm Hg systolic and 90 mm Hg diastolic), hypotension (20 mmHg decrease in blood pressure from baseline, provided this is <100 mm Hg systolic or 60 mm Hg diastolic), bradycardia (a decrease in heart rate of >20 bpm, provided this is less than 60), tachycardia (an increase in heart rate of >20 bpm, provided this >100 bpm)
Arm/Group | Diphenhydramine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/58
Other Adverse Events (participants affected / at risk) | 17/61 | 25/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diphenhydramine (N=61) | Placebo (N=58)
Hypertension (General disorders) | 5 (5) | 3 (3)
Hypotension (Cardiac disorders) | 12 (12) | 22 (22)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0)
Reversal Agent (General disorders) | 0 (0) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT01967433/Prot_SAP_000.pdf